CLINICAL TRIAL: NCT02381158
Title: Nebulized Beclomethasone Dipropionate Improves Respiratory Lung Function in Preschool Children With Recurrent Wheezing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Responsible Party: Principal Investigator, Stefania La Grutta, MD, MD, Istituto per la Ricerca e l'Innovazione Biomedica
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0000573
Record Dates: First submitted 2015-02-12; First posted 2015-03-06 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Wheezing
Keywords: Wheezing; Children
MeSH Terms: conditions — Respiratory Sounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nebulized Beclomethasone dipropionate (Experimental): Nebulized Beclomethasone dipropionate applied for 12 weeks with a dose of 400 µg twice a day (total dose 800 µg).
  Interventions: Drug: Nebulized beclomethasone dipropionate

INTERVENTIONS:
Drug: Nebulized beclomethasone dipropionate — Nebulized beclomethasone dipropionate applied for 12 weeks with a dose of 400 µg twice a day (total dose 800 µg)
  Other Names: BDP

SUMMARY:
This is a single-centre, open label study, aiming to evaluate the efficacy of beclomethasone dipropionate applied for 12 weeks with a dose of 400 µg twice a day (total dose 800 µg nebulized), on airway resistance and reactances (measured with Rint and FOT techniques) in children with recurrent wheezing, aged 2-5 years. In addition, clinic score as frequency of symptoms and exacerbations, will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Informed and subscribed consent before any procedure
* Age range : 2 - ≤5 years
* Male and female patients
* Recurrent wheezing affected ( ≥ 4 episodes in the last 12 months)
* PAI positive (at least one primary and two secondary ):

Primary:

1. one parent with asthma
2. Atopic Dermatitis
3. sensibilisation to air allergen

Secondary:

1. Food sensibilization
2. wheezing also not during the infective episodes
3. eosinophilia (>4%)

Exclusion Criteria:

* story of severe wheeze requiring hospitalization
* treatment with inhaled glucocorticoids during the previous 4 weeks or with oral glucocorticoids in the previous 8 weeks
* structural abnormalities of the lungs (tracheobronchial bronchomalacia, external compressions, etc)
* Persistent infections
* aspiration lung disease (gastroesophageal reflux disease, etc.)
* Cystic fibrosis
* prematurity or bronchopulmonary dysplasia
* Tuberculosis
* primary ciliary dyskinesia
* congenital heart disease
* pulmonary foreign body
* bronchiectasis
* Immunodeficit

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Lung fuction with Rint and FOT | 12 Weeks